CLINICAL TRIAL: NCT02840474
Title: VRC 607-ACTG A5378: A Phase 1, Single Dose Study of the Safety and Virologic Effect of an HIV-1 Specific Broadly Neutralizing Human Monoclonal Antibody, VRC-HIVMAB080-00-AB (VRC01LS) or VRC-HIVMAB075-00-AB (VRC07-523LS), Administered Intravenously to HIV-Infected Adults.
Brief Title: Phase 1, Open-label, Single Dose Study to Examine Safety, Tolerability, Pharmacokinetics and Virologic Impact of VRC01LS or VRC07-523LS in HIV-infected Viremic Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160147; 16-I-0147 (Other: NIH IRB); 30089 (Other: DAIDS)
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Results first posted 2021-02-23 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-12

CONDITIONS: HIV-1
Keywords: HIV Viral Load; Antiviral; CD4 Count; HIV-1 Infection; Broadly Neutralizing Antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: VRC01LS (40 mg/kg) (Experimental): VRC-HIVMAB080-00-AB (VRC01LS) - (40 mg/kg) - administered intravenously (IV) at Day 0
  Interventions: Biological: VRC-HIVMAB080-00-AB
- Part B: VRC07-523LS (40 mg/kg) (Experimental): VRC-HIVMAB075-00-AB (VRC07-523LS) - (40 mg/kg) - administered IV at Day 0
  Interventions: Biological: VRC-HIVMAB075-00-AB

INTERVENTIONS:
Biological: VRC-HIVMAB080-00-AB — VRC01LS is an investigational human monoclonal antibody targeted to the CD4+ binding site of HIV-1.
  Other Names: VRC01LS
  Arms: Part A: VRC01LS (40 mg/kg)
Biological: VRC-HIVMAB075-00-AB — VRC07-523LS is an investigational human monoclonal antibody targeted to the CD4+ binding site of HIV-1.
  Other Names: VRC07-523LS
  Arms: Part B: VRC07-523LS (40 mg/kg)

SUMMARY:
Background:

The human body uses antibodies as one way to help fight infection. VRC01LS and VRC07-523LS are antibodies directed against the HIV virus. Researchers want to see if they are safe and well tolerated. In Part A of the study, the researchers studied VRC01LS. Part A of the study was completed in 2017. In Part B, the researchers studied VRC07-523LS. Depending on which antibody received, researchers studied the amount of VRC01LS or VRC07-523LS in the body and how it changes over time. They evaluated the effect of antibodies on CD4+ (Cluster of Differentiation 4) lymphocyte count and HIV viral load, and checked to see if people who get VRC01LS or VRC07-523LS develop an immune response to it.

Objective:

To see if VRC01LS and VRC07-523LS are safe and well tolerated.

Eligibility:

Adults ages 18-70 who are HIV infected but otherwise healthy.

Design:

Participants received the study drug one time by IV infusion. A needle guided a thin tube into a vein. The study drug mixed with salt water was dripped into the vein over about 30 minutes.

Participants were monitored for 30 minutes after the infusion.

Blood samples were taken at the following times:

* Once before the infusion
* 5 times in the 4 hours after the infusion
* 1 time 24 hours after infusion. Some participants may have had 3 optional blood draws in the time period between 4 and 24 hours.

For 3 days after the infusion, participants recorded their temperature and reactogenicity symptoms in a diary.

There were a total of 23 study visits over 48 weeks. Ten visits were in the first 4 weeks. At all visits, participants answered health questions and gave blood samples.

DETAILED DESCRIPTION:
Study Design:

Open-label, single dose study to examine safety, tolerability, pharmacokinetics and virologic impact of VRC01LS or VRC07-523LS in HIV-infected viremic adults.

Study Hypotheses:

This is the first study of VRC01LS or VRC07-523LS in HIV-infected viremic adults. The primary hypothesis is that both VRC01LS and VRC07-523LS will be safe for intravenous administration to HIV-1-infected adults. The secondary hypothesis is that VRC01LS and VRC07-523LS will be detectable in human sera with a definable half-life.

Product Description:

VRC-HIVMAB080-00-AB (VRC01LS) and VRC-HIVMAB075-00-AB (VRC07-523LS) are human monoclonal antibodies (MAbs) targeted to the CD4+ binding site of HIV-1. Both MAbs are modifications of the VRC01 MAb (which has been shown to be safe and to have antiviral activity in human studies) with the addition of the "LS", a 2-amino acid mutation designed to improve the half-life of the antibody. These MAbs were developed and manufactured by VRC/NIAID/NIH under current Good Manufacturing Practice (cGMP) at the VRC Vaccine Pilot Plant operated under contract by the Vaccine Clinical Materials Program (VCMP), Leidos Biomedical Research, Inc., Frederick, MD. Vials were provided at 100 mg/mL.

Participants:

HIV-1-infected viremic adults; 18-70 years of age.

Study Plan:

This study assessed VRC01LS or VRC07-523LS administered at 40 mg/kg IV in HIV-infected viremic participants. Participants enrolled in one of two parts: Part A (VRC01LS) or Part B (VRC07-523LS). A total of 7 participants were enrolled in Part A and received VRC01LS and a total of 9 participants were enrolled in Part B and received VRC07-523LS. Safety lab samples, HIV viral load, CD4+ lymphocyte count, pharmacokinetic (PK) samples, and blood samples for detection of human anti-VRC01LS antibody (Part A) and human anti-VRC07-523LS antibody (Part B) were drawn at baseline and intervals throughout the study. Participants recorded in a daily diary reactogenicity symptoms for 3 days after study product administration and were queried at each study visit for adverse events. Participants were strongly encouraged to initiate 3-drug anti-retroviral therapy (ART), prescribed by their primary HIV clinician; not study-provided, any time after completing the day 14 study evaluations.

VRC 607/A5378 Study Schema:

* Part: A; Participants: 7; Product: VRC01LS; Administration Schedule (Day 0): 40 mg/kg IV.
* Part: B; Participants: 9; Product: VRC07-523LS; Administration Schedule (Day 0): 40 mg/kg IV.

  * Total Participants: 16

Study Duration:

Participants were followed for 48 weeks after study product administration.

ELIGIBILITY:
INCLUSION CRITERIA:

A participant must meet all of the following criteria:

1. Able and willing to complete the informed consent process.
2. 18-70 years old
3. Available for clinic visits for 48 weeks after study product administration.
4. HIV-1 infected and clinically stable. [Note: Documented HIV-1 infection by HIV enzyme immunoassay (EIA) performed by a Clinical Laboratory Improvement Amendments (CLIA) certified outside lab within 28 days of enrollment is acceptable.]
5. At least one plasma viral load >=500 copies/mL within 28 days of enrollment. A plasma viral load within 28 days and closest to the day of enrollment, that is detectable but not greater than 100,000 copies/mL. [Note: outside laboratory results will be acceptable].
6. A CD4+ count >=350 cells/microliter (mcL) on 2 of 3 consecutive testing occasions (or on 2 of 2 sequential tests) within 28 days prior to enrollment. [Note: outside laboratory results will be acceptable].
7. In general good health as assessed by a study clinician and under the care of a primary health care provider for medical management of HIV infection while participating in the study. Willing to give consent to contact and send laboratory results to the participant's primary health provider.
8. Willing to have blood samples collected, stored indefinitely, and used for various research purposes.
9. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
10. Screening laboratory values within 28 days prior to enrollment must meet the following criteria:

    * Absolute neutrophil count >=800/mcL
    * Platelets >=100,000/mcL
    * Hemoglobin >=10.0 g/dL
    * Creatinine less than or equal to 1.31 mg/dL
    * Alanine aminotransferase (ALT) less than or equal to 2.5 x upper limit of normal (ULN)
    * Negative Hepatitis B Surface Antigen (HBsAg)
    * Undetectable Hepatitis C Viral Load (HCV RNA)

    [Note: Documented negative HBsAg and HCV RNA performed by an outside CLIA certified lab within 28 days of enrollment are acceptable.]

    Female-Specific Criteria:
11. If a woman is sexually active with a male partner and has no history of hysterectomy, tubal ligation, or menopause, she must agree to use either a prescription birth control method or a barrier birth control method from the time of study enrollment until the last study visit, or have a monogamous partner who has had a vasectomy.
12. Negative beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

EXCLUSION CRITERIA:

A participant will be excluded if one or more of the following conditions apply:

1. Previous receipt of humanized or human monoclonal antibody whether licensed or investigational.
2. Prior use of antiretroviral therapy.
3. Ongoing AIDS-related opportunistic infection (including oral thrush).
4. Active drug or alcohol use or dependence in the opinion of the site investigator that would interfere with adherence to study requirements.
5. Any history of a severe allergic reaction, including generalized urticaria, angioedema or anaphylaxis prior to enrollment, that has a reasonable risk of recurrence during the study.
6. Physical finding on examination considered clinically significant.
7. Hypertension that is not well controlled.
8. Weight >115 kg (253 pounds).
9. Breast-feeding.
10. Receipt of any investigational study product within 28 days prior to enrollment.
11. Any other chronic or clinically significant medical condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin R Gaudinski, M.D., Study Chair — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (7):
- United States (6):
  - University of Alabama HIV Clinic Clinical Research Site, AIDS Clinical Trials Group (ACTG), Birmingham, Alabama
  - UCLA CARE Center, AIDS Clinical Trials Group (ACTG), Los Angeles, California
  - Washington University Therapeutics, AIDS Clinical Trials Group (ACTG), St Louis, Missouri
  - University of Cincinnati University Hospital, AIDS Clinical Trials Group (ACTG), Cincinnati, Ohio
  - Ohio State University Clinical Research Site, AIDS Clinical Trials Group (ACTG), Columbus, Ohio
  - Hospital of the University of Pennsylvania Clinical Research Site, AIDS Clinical Trials Group (ACTG), Philadelphia, Pennsylvania
- Puerto Rico AIDS Clinical Trials Unit, AIDS Clinical Trials Group (ACTG), San Juan, PR, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ledgerwood JE, Coates EE, Yamshchikov G, Saunders JG, Holman L, Enama ME, DeZure A, Lynch RM, Gordon I, Plummer S, Hendel CS, Pegu A, Conan-Cibotti M, Sitar S, Bailer RT, Narpala S, McDermott A, Louder M, O'Dell S, Mohan S, Pandey JP, Schwartz RM, Hu Z, Koup RA, Capparelli E, Mascola JR, Graham BS; VRC 602 Study Team. Safety, pharmacokinetics and neutralization of the broadly neutralizing HIV-1 human monoclonal antibody VRC01 in healthy adults. Clin Exp Immunol. 2015 Dec;182(3):289-301. doi: 10.1111/cei.12692. Epub 2015 Sep 24. PMID 26332605
- [Background] Lynch RM, Boritz E, Coates EE, DeZure A, Madden P, Costner P, Enama ME, Plummer S, Holman L, Hendel CS, Gordon I, Casazza J, Conan-Cibotti M, Migueles SA, Tressler R, Bailer RT, McDermott A, Narpala S, O'Dell S, Wolf G, Lifson JD, Freemire BA, Gorelick RJ, Pandey JP, Mohan S, Chomont N, Fromentin R, Chun TW, Fauci AS, Schwartz RM, Koup RA, Douek DC, Hu Z, Capparelli E, Graham BS, Mascola JR, Ledgerwood JE; VRC 601 Study Team. Virologic effects of broadly neutralizing antibody VRC01 administration during chronic HIV-1 infection. Sci Transl Med. 2015 Dec 23;7(319):319ra206. doi: 10.1126/scitranslmed.aad5752. PMID 26702094
- [Background] Ko SY, Pegu A, Rudicell RS, Yang ZY, Joyce MG, Chen X, Wang K, Bao S, Kraemer TD, Rath T, Zeng M, Schmidt SD, Todd JP, Penzak SR, Saunders KO, Nason MC, Haase AT, Rao SS, Blumberg RS, Mascola JR, Nabel GJ. Enhanced neonatal Fc receptor function improves protection against primate SHIV infection. Nature. 2014 Oct 30;514(7524):642-5. doi: 10.1038/nature13612. Epub 2014 Aug 13. PMID 25119033
- [Derived] Happe M, Lynch RM, Fichtenbaum CJ, Heath SL, Koletar SL, Landovitz RJ, Presti RM, Santana-Bagur JL, Tressler RL, Holman LA, Novik L, Roa JC, Rothwell RS, Strom L, Wang J, Hu Z, Conan-Cibotti M, Bhatnagar AM, Dwyer B, Ko SH, Belinky F, Namboodiri AM, Pandey JP, Carroll R, Basappa M, Serebryannyy L, Narpala SR, Lin BC, McDermott AB, Boritz EA, Capparelli EV, Coates EE, Koup RA, Ledgerwood JE, Mascola JR, Chen GL, Tebas P; VRC 607/A5378 Study Team. Virologic effects of broadly neutralizing antibodies VRC01LS and VRC07-523LS on chronic HIV-1 infection. JCI Insight. 2025 Feb 24;10(4):e181496. doi: 10.1172/jci.insight.181496. PMID 39989458
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-I-0147.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant in Part A enrolled in April 2017 and recruitment closed in October 2017. The first participant in Part B enrolled in November 2018 and recruitment closed in February 2019.
Period: Overall Study
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Started | 7 | 9
Received Study Product | 7 | 9
Completed | 6 | 9
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: Population includes all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg) | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Customized [Count of Participants; unit: Participants]
  18-20 years old | 0 | 2 | 2
  21-30 years old | 3 | 4 | 7
  31-40 years old | 1 | 2 | 3
  41-50 years old | 1 | 0 | 1
  51-60 years old | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 5 | 9 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 5 | 1 | 6
  White | 2 | 7 | 9
  Race Unknown/Not Reported | 0 | 1 | 1
  Hispanic/Latino | 0 | 2 | 2
  Non-Hispanic/Latino | 7 | 7 | 14
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 91.2 (22.2) | 81.4 (19.5) | 85.7 (20.6)
HIV Status - positive [Count of Participants; unit: Participants]
  Not on Antiretroviral Treatment | 7 | 9 | 16
  On Antiretroviral Treatment | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms for 3 Days After VRC01LS or VRC07-523LS Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 3 days after the study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0 [November 2014].
Time Frame: 3 days after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) and provided safety data (via diary card) following the administration (N=16).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
Participants
  Pain/Tenderness: None | 7 | 6
  Pain/Tenderness: Mild | 0 | 3
  Pain/Tenderness: Moderate | 0 | 0
  Pain/Tenderness: Severe | 0 | 0
  Bruising: None | 7 | 7
  Bruising: Mild | 0 | 2
  Bruising: Moderate | 0 | 0
  Bruising: Severe | 0 | 0
  Swelling: None | 7 | 9
  Swelling: Mild | 0 | 0
  Swelling: Moderate | 0 | 0
  Swelling: Severe | 0 | 0
  Redness: None | 7 | 9
  Redness: Mild | 0 | 0
  Redness: Moderate | 0 | 0
  Redness: Severe | 0 | 0
  Pruritus: None | 7 | 9
  Pruritus: Mild | 0 | 0
  Pruritus: Moderate | 0 | 0
  Pruritus: Severe | 0 | 0
  Any Local Symptom: None | 7 | 6
  Any Local Symptom: Mild | 0 | 3
  Any Local Symptom: Moderate | 0 | 0
  Any Local Symptom: Severe | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms for 3 Days After VRC01LS or VRC07-523LS Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 3 days after the study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0 [November 2014].
Time Frame: 3 days after study product administration
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
Participants
  Malaise: None | 7 | 7
  Malaise: Mild | 0 | 2
  Malaise: Moderate | 0 | 0
  Malaise: Severe | 0 | 0
  Myalgia: None | 7 | 8
  Myalgia: Mild | 0 | 1
  Myalgia: Moderate | 0 | 0
  Myalgia: Severe | 0 | 0
  Headache: None | 6 | 8
  Headache: Mild | 1 | 1
  Headache: Moderate | 0 | 0
  Headache: Severe | 0 | 0
  Chills: None | 6 | 9
  Chills: Mild | 1 | 0
  Chills: Moderate | 0 | 0
  Chills: Severe | 0 | 0
  Nausea: None | 6 | 9
  Nausea: Mild | 1 | 0
  Nausea: Moderate | 0 | 0
  Nausea: Severe | 0 | 0
  Temperature: None | 7 | 9
  Temperature: Mild | 0 | 0
  Temperature: Moderate | 0 | 0
  Temperature: Severe | 0 | 0
  Joint Pain: None | 7 | 9
  Joint Pain: Mild | 0 | 0
  Joint Pain: Moderate | 0 | 0
  Joint Pain: Severe | 0 | 0
  Any Systemic Symptom: None | 6 | 7
  Any Systemic Symptom: Mild | 1 | 2
  Any Systemic Symptom: Moderate | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety
Description: Any abnormal laboratory results recorded as unsolicited AEs are summarized. Labs included hematology (hemoglobin, hematocrit, mean corpuscular volume (MCV), platelets, white blood cell (WBC) and red blood cell (RBC) counts, and neutrophil, lymphocyte, monocyte, eosinophil and basophil percents and counts) and chemistry (alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and creatinine). Complete blood count (CBC) and platelet results were collected at screening, Day 0 prior to study product administration (baseline), and Days 2 and 7, Weeks 2-8, 12, 16, 20, 24, 36 and 48 after product administration. Creatinine, ALT, AST and ALP results were collected at screening, baseline, and Days 2 and 7, Weeks 2, 4, 12, 24, 36 and 48 after product administration. Institutional laboratory normal ranges as well as the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.0 [November 2014] were used.
Time Frame: Through 48 weeks after study product administration
Population: Population included all enrolled participants who had laboratory results available at any study visit post baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
Participants
  ALT | 0 | 2
  AST | 0 | 2
  Neutrophil Count | 0 | 1

4. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs)
Description: Unsolicited AEs and attribution assessments were recorded in the study database from receipt of the study product administration through the visit scheduled for 56 days (or 8 weeks) after study product administration. At other time periods greater than 56 days (or 8 weeks) after the study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module), and new chronic medical conditions that required ongoing medical management were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Through 56 days after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
Participants
  Related to Study Product | 0 | 2
  Unrelated to Study Product | 2 | 6

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: SAEs were recorded from receipt of the study product administration through the last expected study visit at Week 48. The relationship between a SAE and the study product was assessed by the investigator on the basis of his or her clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Through 48 weeks after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
Participants
  Related to Study Product | 0 | 0
  Unrelated to Study Product | 1 | 0

6. Secondary Outcome: Area Under the Curve For the Last Study Visit (AUC(Last))
Description: The AUC(last) represents the area under the curve (AUC) from zero (dosing) to the time of the last measurable drug concentration at the last study visit after study product administration; it is determined based on the summary PK curve for each study group.
  Serum samples were collected pre-infusion (baseline), end of infusion (0h), 30 min, 1 hr-4 hr, 24 hr, 48 hr and Days 7, 14, 21, 28, 35, 42, 49, 56, 84, 112, 140, 168, 252 and 336 (Week 48) post-infusion.
Time Frame: Administration (0h) to 48 weeks after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Mean (Standard Deviation); unit: µg*d/mL
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
µg*d/mL | 34280 (2796) | 17967 (4563)

7. Secondary Outcome: Clearance Rate of VRC01LS or VRC07-523LS Administered at 40 mg/kg IV
Description: Rate of study product elimination divided by the plasma concentration; determined based on the summary PK curve for each study group. Serum samples were collected pre-infusion (baseline), end of infusion (0h), 30 min, 1 hr-4 hr, 24 hr, 48 hr and Days 7, 14, 21, 28, 35, 42, 49, 56, 84, 112, 140, 168, 252 and 336 (Week 48) post-infusion.
Time Frame: Administration (0h) to 48 weeks after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Mean (Standard Deviation); unit: mL/d
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
mL/d | 104.3 (21.4) | 188.7 (55.8)

8. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of VRC01LS or VRC07-523LS Administered at 40 mg/kg IV
Description: Cmax is the peak serum concentration that the study product achieves after it has been administered; it is determined as a maximum value on the summary pharmacokinetic (PK) curve for each study group. Serum samples were collected pre-infusion (baseline), end of infusion (0h), 30 min, 1 hr-4 hr, 24 hr, 48 hr and Days 7, 14, 21, 28, 35, 42, 49, 56, 84, 112, 140, 168, 252 and 336 (Week 48) post-infusion.
Time Frame: Through 48 weeks after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
mcg/mL | 1566.3 (315.6) | 1295.2 (375.9)

9. Secondary Outcome: Half-life (T1/2) of VRC01LS or VRC07-523LS Administered at 40 mg/kg IV
Description: Half-life (T1/2) is the time required for half of the study product to be eliminated from the serum. Serum samples were collected pre-infusion (baseline), end of infusion (0h), 30 min, 1 hr-4 hr, 24 hr, 48 hr and Days 7, 14, 21, 28, 35, 42, 49, 56, 84, 112, 140, 168, 252 and 336 (Week 48) post-infusion.
Time Frame: Through 48 weeks after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
Days | 47.3 (8.4) | 56.5 (13.2)

10. Secondary Outcome: Mean Serum Concentration of VRC01LS or VRC07-523LS Administered at 40 mg/kg IV
Description: The mean of individual subject serum concentrations by administered study group. Serum samples were collected pre-infusion (baseline), end of infusion (0h), 30 min, 1 hr-4 hr, 24 hr, 48 hr and Days 7, 14, 21, 28, 35, 42, 49, 56 and 84 post-infusion.
Time Frame: Day 28 and Day 84 after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
mcg/mL
  Concentration at Day 28 | 336.4 (68.6) | 162.6 (42.7)
  Concentration at Day 84 | 136.2 (21.9) | 60.7 (20.8)

11. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of VRC01LS or VRC07-523LS Administered at 40 mg/kg IV
Description: Tmax is the time it takes to reach Cmax of study product after it has been administered; it is determined based on the summary PK curve for each study group.
  Serum samples were collected pre-infusion (baseline), end of infusion (0h), 30 min, 1 hr-4 hr, 24 hr, 48 hr and Days 7, 14, 21, 28, 35, 42, 49, 56, 84, 112, 140, 168, 252 and 336 (Week 48) post-infusion.
Time Frame: Through 48 weeks after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
Days | 0.07 (0.06) | 0.06 (0.05)

12. Secondary Outcome: Number of Participants Who Produced Anti-drug Antibodies to VRC01LS or VRC07-523LS Administered at 40 mg/kg IV
Description: Presence of anti-drug antibodies to VRC01LS or VRC07-523LS was evaluated.
Time Frame: Day 28 and Day 56 after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16) and had serum samples collected at Day 28 and Day 56 post administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
Participants
  Day 28 (Week 4): Participants with Anti-Drug Antibodies | 0 | 0
  Day 56 (Week 8): Participants with Anti-Drug Antibodies | 0 | 0
  Total number of Participants with Anti-Drug Antibodies | 0 | 0

13. Secondary Outcome: Log10 Change in Viral Load (VL) From Baseline to Nadir (Lowest Detectable Value) Prior to Antiretroviral Therapy (ART) Initiation
Description: Baseline VL (log10) was the average of VL (log10) at the enrollment and pre-administration study visits. Nadir (lowest detectable) values were calculated pre-ART. For participants who didn't get ART, nadir was calculated as the minimum VL (log10) from baseline through the last visit.
Time Frame: Baseline through 48 weeks after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
log10 copies/mL
  Baseline VL | 3.6 (0.9) | 4.5 (0.4)
  Nadir VL (prior to ART) | 2.6 (1.5) | 2.8 (0.5)
  Decline in VL from Baseline to Nadir (prior to ART) | 1.0 (1.1) | 1.7 (0.7)

14. Secondary Outcome: Day of Nadir (Lowest Detectable) VL Prior to ART Initiation
Description: Nadir values were calculated pre-ART. For participants who didn't get ART, nadir was calculated from baseline through the last visit.
Time Frame: Baseline through 48 weeks after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
Days | 45.2 (91.8) | 9.0 (4.1)

15. Secondary Outcome: Overall Change in CD4+ Lymphocyte Count From Baseline to Peak Prior to ART Initiation
Description: The pre-administration study visit was considered the baseline visit. Peak values were calculated pre-ART. For participants who didn't get ART, peak was calculated as the maximum CD4+ lymphocyte counts from baseline through the last visit.
Time Frame: Baseline through 48 weeks after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Mean (Standard Deviation); unit: cells/mcL
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
cells/mcL
  Baseline CD4+ Count | 540.1 (138.6) | 566.9 (165.1)
  Peak CD4+ Count post baseline (prior to ART) | 668.4 (236.4) | 719.1 (233.9)
  Increase in CD4+ Count from Baseline to Peak (prior to ART) | 128.3 (171.1) | 152.2 (160.8)

16. Secondary Outcome: Day of Peak CD4+ Lymphocyte Count Prior to ART Initiation
Description: Peak values were calculated pre-ART. For participants who didn't get ART, peak was calculated as the maximum CD4+ counts from baseline through the last visit.
Time Frame: Baseline through 48 weeks after study product administration
Population: Population included all enrolled participants who received study product (VRC01LS or VRC07-523LS) (N=16).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
Number analyzed (Participants) | 7 | 9
Days | 59.0 (86.3) | 11.7 (6.1)

ADVERSE EVENTS:
Time Frame: Solicited adverse events (AEs) were reported for 3 days after study product administration. Unsolicited AEs were recorded from receipt of the study product through the visit scheduled 56 days (or 8 weeks) after administration. At other time periods greater than 56 days after product administration, only serious AEs and new chronic medical conditions that required ongoing medical management were recorded through the last study visit.
Description: All AEs recorded on the study were reported. Solicited AEs collected through systematic assessment and unsolicited AEs collected through non-systematic assessment are reported for participants who received study product and had safety data collected following the product administration. Data represent the number and percentage of participants experiencing the event. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Part A: VRC01LS (40 mg/kg) | Part B: VRC07-523LS (40 mg/kg)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/9
Other Adverse Events (participants affected / at risk) | 2/7 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: VRC01LS (40 mg/kg) (N=7) | Part B: VRC07-523LS (40 mg/kg) (N=9)
Gout (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: VRC01LS (40 mg/kg) (N=7) | Part B: VRC07-523LS (40 mg/kg) (N=9)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Eye pain (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Infusion site paraesthesia (General disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood pressure diastolic increased (Investigations) | 0 | 2
Blood pressure systolic increased (Investigations) | 0 | 4
Neutrophil count decreased (Investigations) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Administration Site Pain/Tenderness (General disorders) | 0 | 3
Administration Site Bruising (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT02840474/Prot_SAP_ICF_000.pdf